CLINICAL TRIAL: NCT02946008
Title: A Phase I Trial of Neoadjuvant Stereotactic Body Radiotherapy Prior to Radical Prostatectomy for High Risk Prostate Cancer
Brief Title: Neoadjuvant Stereotactic Body Radiotherapy Prior to Radical Prostatectomy for High Risk Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2016.106; HUM00120414 (Other: University of Michigan)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SBRT (Experimental): Stereotactic Body Radiation Therapy (SBRT) will be delivered over 5 treatment sessions for approximately 1.5 weeks total.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Procedure: Radical Prostatectomy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Delivered over 5 treatment sessions for approximately 1.5 weeks total.
Procedure: Radical Prostatectomy — Open, laparoscopic, or robotic radical prostatectomy and pelvic lymph node dissection to remove the prostate, seminal vesicles, and pelvic lymph nodes.

SUMMARY:
This is a single-arm prospective non-randomized, non-blinded trial to assess the safety of neoadjuvant stereotactic body radiation therapy (SBRT) before surgery in high risk prostate cancer patients.

Radiation therapy will be delivered over 5 treatment sessions for approximately 1.5 weeks total.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have biopsy-confirmed adenocarcinoma of the prostate.
* Subjects must have a negative bone scan.
* Subjects must have one of the following risk factors:
* PSA ≥20 and/or
* Gleason score ≥8 and/or
* Clinical or radiographic stage ≥T3a per AJCC (American Joint Committee on Cancer) 7th Edition Staging Manual and/or
* Radiographic pelvic lymph node positive disease and/or
* At least two out of four of the following: PSA (Prostate Specific Antigen) 10-19.9, GS (Gleason Score) = 3+4, clinical stage = T2b/T2c, ≥50% positive biopsy cores.
* Subjects must freely sign informed consent to enroll in the study.
* Subjects must be medically fit to undergo surgery determined by the PI.
* Age ≥ 18
* KPS Karnofsky Performance Status (performance status is an attempt to quantify cancer patients' general well-being and activities of daily life, scores range from 0 to 100 where 100 represents perfect health and 0 represents death): ≥70.
* No prior invasive malignancy in the past 3-years, except non-melanomatous skin cancer unless disease free for a minimum of 2 years. Carcinoma in-situ of the bladder or head and neck region is permissible.
* Subjects must not have had prior pelvic radiation therapy,
* Subjects must not have had prior androgen deprivation therapy in the past 6 months.

Exclusion Criteria:

* Metastatic disease as demonstrated by bone scan, CT scan or MRI (Magnetic Resonance Imaging) of the pelvis, or chest x-ray.
* Declared high-risk for anesthesia by attending anesthesiologist, cardiologist, or other physician.
* History of prior pelvic radiation therapy.
* History of androgen deprivation therapy within the past 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Neoadjuvant SBRT | 6-week post-prostatectomy
  The MTD is defined as the SBRT dose that with radical prostatectomy induces dose-limiting toxicity in 28% of subjects or less.

SECONDARY OUTCOMES:
Incidence of Urinary Incontinence | up to one year post treatment
  Urinary incontinence will be scored according to Common Toxicity Criteria for Adverse Events (CTCAE) v.4.0 (Grade 1 = Occasional, Grade 2 = Spontaneous, pads indicated, Grade 3 = Intervention indicated)
Incidence of Urinary Stricture | up to one year post treatment
  Urinary stricture, according to Common Toxicity Criteria for Adverse Events (CTCAE) v.4.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening, Grade 5 = death.)
Incidence of Urinary Bother | up to one year post treatment
  Urinary bother, according to Common Toxicity Criteria for Adverse Events (CTCAE) v.4.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening, Grade 5 = death.)
Rectal Toxicity | up to one year post treatment
  Rectal Toxicity, according to Common Toxicity Criteria for Adverse Events (CTCAE) v.4.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening, Grade 5 = death.)
Number of Patients with Positive Surgical Margins | 4-10 weeks post radiation therapy
  Surgical specimens will be evaluated by the study pathologist to determine rate of margin positivity.
Number of Patients with Extracapsular Extension | 4-10 weeks post radiation therapy
  Surgical specimens will be evaluated by the study pathologist to determine rate of extracapsular extension.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Spratt, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hammer L, Jiang R, Hearn J, Lashbrook J, Mitchell A, Daignault-Newton S, Dess RT, Jackson WC, Reichert Z, Alumkal JJ, Kaffenberger S, George A, Montgomery J, Salami SS, Morgan TM, Miller D, Wittman D, Hollenbeck B, Mehra R, Davenport MS, Sun Y, Schipper M, Palapattu G, Spratt DE. A Phase I Trial of Neoadjuvant Stereotactic Body Radiotherapy Prior to Radical Prostatectomy for Locally Advanced Prostate Cancer. Int J Radiat Oncol Biol Phys. 2023 Jan 1;115(1):132-141. doi: 10.1016/j.ijrobp.2022.07.016. Epub 2022 Jul 22. PMID 35878714